CLINICAL TRIAL: NCT03087006
Title: Automatic Self Transcending Meditation (ASTM) Plus Treatment As Usual (TAU) Versus TAU Alone in Patients With Dry Eye Disease (DED): a Single Blind Randomized Controlled Longitudinal Study
Brief Title: Automatic Self Transcending Meditation (ASTM) in Patients With Dry Eye Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Monali Malvankar, Assistant Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 108461
Record Dates: First submitted 2017-03-10; First posted 2017-03-22 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Eye Diseases; Quality of Life; Depression; Anxiety
MeSH Terms: conditions — Eye Diseases; Depression; Anxiety Disorders | interventions — Meditation; Therapeutics; Primary Health Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Automatic Self Transcending Meditation (Active Comparator): Automatic Self Transcending Meditation (ASTM) may help with depression, anxiety, stress, PTSD, and may have a positive impact on quality of life of participants diagnosed with dry eye disease. ASTM is a class of meditation that helps quiet the mind and induces physiological and mental relaxation whilst the eyes are shut. It utilizes a specific sound value (mantra) to draw attention inward and permit the mind to experience a restful but alert state of consciousness.
  Interventions: Other: Automatic Self Transcending Meditation (ASTM)
- Treatment as Usual (TAU) (Placebo Comparator): Participants continue to receive treatment as usual including dry eye disease medications.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Other: Automatic Self Transcending Meditation (ASTM) — Automatic Self Transcending Meditation (ASTM) is a class of meditation that helps quiet the mind. Research suggests that ASTM helps reduce depression, anxiety, stress, and may improve health related quality of life. Further, ASTM is easier to learn and to teach.
  Other Names: Meditation
  Arms: Automatic Self Transcending Meditation
Other: Treatment as Usual — Usual Care includes usual care of the participants including dry eye disease medications
  Other Names: Primary Care
  Arms: Treatment as Usual (TAU)

SUMMARY:
Patients with dry eye disease (DED) will be randomized to Automatic Self Transcending Meditation (ASTM) plus Treatment as Usual (TAU) or TAU alone to assess changes in Health-related quality of life (HRQoL). HRQoL is a vital construct focusing on impact of health on quality of life. HRQoL data is used in economic evaluations, a component of health economics that compares the cost and consequences of alternative courses of action. This helps policy-makers make complex financial decisions. Along with HRQoL we will measure changes in extent of depression as well as anxiety. Previously published data lacks information of HRQoL in patients with DED. Through this study we shall attempt to correlate HRQoL in this population and assess if ASTM confers changes in HRQoL along with depressive and anxiety symptoms.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE: Dry eye disease (DED) may degrade vision that can interfere with daily activities including reading, driving, and viewing computer screen. Further, DED is associated with decreased productivity, absenteeism from work, depression, post-traumatic stress disorder (PTSD), and have an adverse impact on patient's quality of life. A category of meditation called Automatic Self Transcending Meditation (ASTM) may help with depression, PTSD, and may have a positive impact on quality of life of participants diagnosed with DED. ASTM is a class of meditation that helps quiet the mind and induces physiological and mental relaxation whilst the eyes are shut. It utilizes a specific sound value (mantra) to draw attention inward and permit the mind to experience a restful but alert state of consciousness. We will offer patients a specific standardized form of ASTM called Sahaj Samadhi Meditation. In this study, we shall measure HRQoL of patients with DED in both ASTM and no intervention arms. HRQoL is an essential measure of quality of life related to health; it helps physician identify hidden morbidities in clinical care as well as improves patient-physician communications. However, majority of current ophthalmic literature describes changes in clinical variables with any intervention whilst lacking information on HRQoL. The reason for lack of HRQoL data in published ophthalmic literature is likely because it is difficult and cumbersome to estimate. Additionally, it is unfortunate that many clinicians severely underestimate the added value of HRQoL measurement in routine clinical practice. We think there is a high necessity to assess if there is an association between HRQoL and routinely measured clinical data. A primary purpose of this study is to assess if ASTM confers beneficial effects on HRQoL of DED patients compared to a no intervention arm. Additionally, we will assess changes, if any, that ASTM confers on self-reported depression and anxiety symptoms as a secondary outcome measure. PRIMARY HYPOTHESIS: We hypothesize that in patients with DED ASTM + TAU will lead to significant improvement in HRQoL compared to TAU alone from baseline to 24 weeks after the initial ASTM training. SECONDARY HYPOTHESES: We hypothesize that in patients with DED 1) HRQoL is associated with regularly measured clinical variables 2) ASTM+TAU leads to significant improvement in depression and anxiety symptoms at 24 weeks compared to TAU alone 3) The beneficial effects of ASTM on all studied variables will be sustained at 24 weeks post intervention. STUDY DESIGN: We plan to conduct a single-center, single blind longitudinal randomized controlled trial. Research participants will be 256 men and women (128 in each group). STUDY RECRUITMENT: Potential participants with mild to severe DED between 18 - 75 years of age will be screened - from the office practice of Dr. Mather as per inclusion and exclusion criteria - by Dr. Mather at the Ivey Eye Institute, London, ON. Letter of information (LOI) will be given to potential participants. An ophthalmic examination - offered as a routine care - for each potential participant (i.e., measuring best-corrected Snellen visual acuity (VA) and pinhole acuities) will be conducted. QUESTIONNAIRE: Patients will undergo a standardized interview performed by a trained interviewer to measure HRQoL using the time trade-off method (TTO) in which potential participants will be asked couple of questions about their quality of life such as 1) how long you expect to live? and 2) how many of those remaining years of life, if any, you would be willing to trade in return for a treatment permitting your current vision in each eye to be transformed to permanent perfect vision (20/20) bilaterally?. During the first office visit only, also a screening visit, in the interview, patients will be asked demographic questions including age, gender, and associated medical conditions, such as concurrent ocular conditions, ocular disease other than DED, previous ocular surgery, inflammation, intraoperative complications, preoperative ocular pathology, chronic pain, general diseases that could affect the immune system, and actual infection. In addition, patients will be asked about co-morbidities such as, whether they have high blood pressure, diabetes, arthritis, heart condition, stroke, and other non-ocular medical conditions. Further, the following self-rated scales will be administered at the first office visit: TTO, Visual Function Questionnaire (VFQ-25), the Patient Health Questionnaire (PHQ-9), Generalized Anxiety Disorder (GAD-7), Canadian Dry Eye Assessment (CDEA), Ocular Surface Disease Index (OSDI), and SPEED Dry Eye Questionnaire. RANDOMIZATION: Participants will be randomized to either ASTM + TAU or TAU alone equally (1:1) using computer generated randomization numbers available at random.org. Concealment of randomization will be ensured by independent staff performing randomization using a third-party web based provider (http://www.sealedenvelope.com/). Computerized randomization will occur from the clinic of Dr. Mather, Ivey Eye Institute in St. Joseph's Hospital, London, Ontario. A telephone number will be available for study concerns/queries. Pre-randomized information will be stored using unique de-identifiers and downloaded on a secure database. It will not be possible to blind participants to intervention status. Outcome assessors and investigators will be blinded to treatment. It will not be possible to blind participants or staff providing treatment to the intervention status. TREATMENT ARMS: 1. Automatic Self-Transcending meditation (ASTM): Following the initial measurements (common to both ASTM and control group), participants in the ASTM group will undergo ASTM training in groups of 10 by certified teachers under the supervision of one of the study collaborator at a room in St. Joseph's Hospital or at the Ivey Eye Institute, 268 Grosvenor Street, London, ON. This involves participating in four, 90-120 minute sessions each of four consecutive days. This will be followed by weekly 60 minute follow up sessions for 4 weeks, biweekly sessions for weeks 5- 12 weeks and monthly follow-up session for 13-24 weeks. Participants will be required to attend 75% of weekly, bi-weekly, monthly follow-up sessions. In addition, participants will be asked to practice ASTM at home for 20 minutes twice daily over the study period (24 weeks). Participants will be asked to log practice frequency and any other noteworthy observations in the log sheet provided to them. Further, the following self-rated scales will be administered by a trained rater at the fourth ASTM session (week 0) as well as at weeks 4, 8, 12, and 24: TTO, VFQ-25, PHQ-9, GAD-7, CDEA, OSDI, and SPEED Dry Eye Questionnaire. CONTROL INTERVENTION: Participants randomized to control arm (Treatment as Usual, TAU) will continue to receive their treatment as usual including DED medications. They will follow assessment and study procedures as listed below. The following self-rated scales will be administered by a trained rater at weeks 0, 4, 8, 12, and 24: TTO, VFQ-25, PHQ-9, GAD-7, CDEA, OSDI, and SPEED Dry Eye Questionnaire. Following a duration of week 24 into the study participants in TAU arm will also be offered the opportunity to learn ASTM. No study procedures will be applied or any other information collected during this period. STUDY RECRUITMENT: We anticipate to recruit participants at a rate of at least 2 participants/week over a period of 128 weeks allowing attainment of sample size of n=256. There is no obligation for the participants to take part in the study; all participation is voluntary. VARIABLE SPECIFICATION: Dependent variable: A dependent variable is created based on the HRQoL, an interval scale variable taking values between 0.0 and 1.0. Independent variables: Visual acuity in a better-seeing eye, patients' demographic characteristics, including age, gender, and associated medical conditions are the independent variables. Patients' demographic characteristics, including age, are considered as continuous variables. Gender is categorized as male and female and associated medical conditions are categorized as "current medical conditions," which includes concurrent ocular conditions, inflammation; "other diseases," which includes ocular diseases other than DED, chronic pain, general diseases that could affect the immune system, and actual infection; and "medical history," which includes previous ocular surgery, preoperative ocular pathology, and intraoperative complications. Data Grouping: Based on BCVA, study participants will be grouped to visual acuity in better seeing eye (group 1, 20/20 to 20/50; group 2, 20/60 to 20/100; group 3, 20/200 to no light perception). Better seeing will be used since a correlation has been shown between utility score and better seeing eye. These 3 groups were chosen since group 1 represents legal driving vision in Canada, group 2 represents moderate visual acuity loss, and group 3 represents legal blindness. DATA ANALYSIS: As has been done in many other studies, HRQoL will be calculated by dividing the number of years a patient is willing to trade in return for improved quality of life by the estimated numbers of years of remaining life subtracted by 1.0 as given below: HRQoL(U)=1-(number of years a patient is willing to trade in return for improved quality of life)/(estimated number of years of remaining life). Mean, standard deviation, and 95% confidence interval for continuous variables such as utility value, will be calculated. For categorical variables, visual acuity in the better-seeing eye, gender, and associated medical conditions, proportions will be calculated. The chi-square test statistic for independence will be used to compare unwillingness to trade time in TTO. The unpaired, two-tailed Student t-test will be used to evaluate the effect of visual acuity in the better eye in four groups and gender on mean of time trade-off utility values. Non-response issues: Non-respondent patients' characteristics will be compared with respondent patients,' and if they do not appear to be statistically significantly different, then these results will be generalized to the sample and population. Data will be analyzed using STATA Software (Version 15.0). The unit of analysis is the HRQoL. Univariate and bivariate analysis will be performed for each independent variable against the dependent variable to elicit the impact of each factor on the pattern of HRQoL without adjusting for the effect of other variables. Models will be deemed statistically significant if they are associated with a significant F value (p < 0.01) and if they explain over 15% variability of the dependent variable. Only those independent variables that are statistically significantly associated with the HRQoL (p < 0.05) will be used for model construction. Since the dependent variable is continuous, we plan to use a non-linear regression model to assess the effect of each independent variable on the dependent variable, while controlling for the confounders. Multicollinearity, high correlation between independent variables, and interaction effects will be evaluated for the model. VALIDATION ANALYSIS: Validation will be performed on the developed regression model. The collected data will be divided into two portions: one portion, called the "main data," will contain 80% of the samples of the total collected utility values and its associated data; the other portion, called the "test data," will contain the remaining 20%. Validation will be done using test data but having the same coefficient values as the main data to calculate the percentage of correct cases. Similar regression analysis as described above will be performed for vision score measured by VFQ-25, depression score by PHQ-9, anxiety score by GAD-7, CDEA score, OSDI score, and SPEED score.

ELIGIBILITY:
Inclusion Criteria:

* dry eye disease suspects or have mild to severe dry eye disease
* at least between 18 to 75 years of age
* deemed competent such as no language issues or communication barriers, no self-reported or physician diagnosed mental health disorder besides having depressive and anxiety symptoms
* have sufficient hearing to be able to follow verbal instructions and able to sit without physical discomfort for 30 minutes
* willing and able to attend 4 initial ASTM training sessions and at least 80% of follow up sessions
* willing to dedicate 20 minutes twice per day to ASTM practice at their own home.

Exclusion Criteria:

* actively suicidal as per self-report (scoring 2 or more on item 9 of the PHQ-9) or on assessment by the physician
* they are currently participating in other similar studies
* currently practicing any type of formal meditation techniques regularly
* unable or unwilling to answer survey questions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Health-related quality of life (HRQoL) | First office visit, Week 0, 4, 6, 8, 12, and 24
  HRQoL is an essential measure of quality of life related to health; it helps physician identify hidden morbidity in clinical care as well as improves patient-physician communications. HRQoL will be measured using time trade-off questionnaire.

SECONDARY OUTCOMES:
Visual Function Score | First office visit, Week 0, 4, 6, 8, 12, and 24
  Visual Function score will be measured using Visual Function Questionnaire (VFQ-25).
Depression | First office visit, Week 0, 4, 6, 8, 12, and 24
  Depression is a feeling of severe despondency and dejection. Depression will be measured using the Patient Health Questionnaire (PHQ-9).
Anxiety | First office visit, Week 0, 4, 6, 8, 12, and 24
  Anxiety will be measured using Generalized Anxiety Disorder (GAD-7)
Dry Eye Assesment | First office visit, Week 0, 4, 6, 8, 12, and 24
  Dry Eye will be assessed using Canadian Dry Eye Assessment (CDEA), Ocular Surface Disease Index (OSDI), SPEED Dry Eye Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Monali Malvankar, PhD, Principal Investigator — Western University, Canada
Locations (1):
- St. Joseph's Hospital, Ivey Eye Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
De-identified IPD collected in this study will not be available to other researchers (e.g. outside the primary research group). Because the primary research group has the necessary expertise to conduct analysis and do not need any outside help.

REFERENCES:
- [Background] Schein OD, Munoz B, Tielsch JM, Bandeen-Roche K, West S. Prevalence of dry eye among the elderly. Am J Ophthalmol. 1997 Dec;124(6):723-8. doi: 10.1016/s0002-9394(14)71688-5. PMID 9402817
- [Background] Schaumberg DA, Dana R, Buring JE, Sullivan DA. Prevalence of dry eye disease among US men: estimates from the Physicians' Health Studies. Arch Ophthalmol. 2009 Jun;127(6):763-8. doi: 10.1001/archophthalmol.2009.103. PMID 19506195
- [Background] Schaumberg DA, Sullivan DA, Buring JE, Dana MR. Prevalence of dry eye syndrome among US women. Am J Ophthalmol. 2003 Aug;136(2):318-26. doi: 10.1016/s0002-9394(03)00218-6. PMID 12888056
- [Background] Yu J, Asche CV, Fairchild CJ. The economic burden of dry eye disease in the United States: a decision tree analysis. Cornea. 2011 Apr;30(4):379-87. doi: 10.1097/ICO.0b013e3181f7f363. PMID 21045640
- [Background] Wan KH, Chen LJ, Young AL. Depression and anxiety in dry eye disease: a systematic review and meta-analysis. Eye (Lond). 2016 Dec;30(12):1558-1567. doi: 10.1038/eye.2016.186. Epub 2016 Aug 12. PMID 27518547
- [Background] Burns JL., Lee RM, Brown LJ. The effect of meditation on self-reported measures of stress, anxiety, depression, and perfectionism in a college population. Journal of College Student Psychotherapy 25(2): 132-144, 2011.
- [Background] Elder C, Nidich S, Moriarty F, Nidich R. Effect of transcendental meditation on employee stress, depression, and burnout: a randomized controlled study. Perm J. 2014 Winter;18(1):19-23. doi: 10.7812/TPP/13-102. PMID 24626068